CLINICAL TRIAL: NCT02325687
Title: A Pilot Study of Biomarkers in Obstructive Sleep Apnea (OSA): Is There a Correlation Between Cerebrospinal Fluid and Serum Markers of Inflammation in OSA?
Brief Title: A Pilot Study of Biomarkers in Obstructive Sleep Apnea
Acronym: Cytokine OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-100
Record Dates: First submitted 2014-12-10; First posted 2014-12-25 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Arthroplasty, Replacement, Knee; Cerebrospinal Fluid; Inflammation; TNF-alpha; Interleukin-6 (IL-6); Interleukin-8 (IL-8); Interleukin-10 (IL-10); Cytokines; Neurotrophins; BDNF; Beta-NGF; Proteomic Analysis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Inflammation; Pain Insensitivity, Congenital | interventions — Spinal Puncture; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treated OSA (CPAP-compliant) (Experimental): Treated OSA patients will have previously been diagnosed with OSA, and are currently CPAP-compliant. CPAP compliance is defined by daily use of a CPAP machine for at least 4 hours. We will determine if patients are CPAP-compliant by looking at their medical records and pre-operative assessments, as well as directly verifying compliance with the patient.
  Intervention: Lumbar Puncture (Standard-of-Care)
  Interventions: Procedure: Lumbar Puncture (Standard-of-Care)
- Untreated OSA (non-CPAP-compliant) (Experimental): Patients in the untreated OSA group will have previously been diagnosed with OSA, but for some reason do not use a CPAP machine every night. We will determine if patients are CPAP-compliant by looking at their medical records and pre-operative assessments, as well as directly verifying compliance with the patient.
  Intervention: Lumbar Puncture (Standard-of-Care)
  Interventions: Procedure: Lumbar Puncture (Standard-of-Care)
- Control (No suspicion of OSA) (Experimental): Patients in the control group will not have previously been diagnosed with OSA, and are currently not at high risk. We will determine overall risk for OSA using the STOP-BANG questionnaire. Patients with a STOP-BANG score <3 are considered to have minimal risk for OSA and will be included in the control group.
  Intervention: Lumbar Puncture (Standard-of-Care)
  Interventions: Procedure: Lumbar Puncture (Standard-of-Care)

INTERVENTIONS:
Procedure: Lumbar Puncture (Standard-of-Care) — All study patients will have previously consented to undergo either spinal or spinal-epidural anesthesia. Patients will undergo their planned spinal or combined spinal-epidural placement in the OR. At the time of confirmation of placement of the spinal needle (positive CSF flow), 5 mL CSF will be collected and stored. CSF will be drawn using a standard 25g or 27g needle commonly used for anesthesia. The volume of CSF removed will be replaced with 4 cc local anesthetic (1.5% mepivacaine for spinal anesthesia).

SUMMARY:
Obstructive sleep apnea (OSA) is common and is a risk factor for postoperative complications, including respiratory and cardiac events and delirium. Despite this risk, however, there are currently no accepted biomarkers that can predict poor outcomes, making it unclear to see which patients will have complications after surgery, and who might need prolonged monitoring or an extended hospital stay. An improved understanding of the pathophysiology of OSA is required to identify potential biomarkers for outcomes after surgery, as well as to develop new treatments. The aim of this pilot study is to identify serum and cerebrospinal (CSF) biomarkers associated with obstructive sleep apnea (OSA). The presence of cytokines and neurotrophins will be determined and quantified in both patients with OSA and in controls. The CSF samples will additionally be analyzed by proteomic methods to identify potential biomarkers with significantly different levels present in patients with and without OSA. The working hypothesis is that OSA patients who are non-CPAP-compliant will have higher levels of circulating cytokines and lower levels of circulating neurotrophins in serum and CSF, compared to patients who are CPAP-compliant and/or controls.

DETAILED DESCRIPTION:
It is being increasingly understood that OSA represents an inflammatory state, with multiple studies showing increased levels of circulating cytokines, possibly providing the link between OSA and cardiovascular/pulmonary morbidity. In support of this, use of CPAP therapy is associated with a reduction in the levels of circulating cytokines in patients with OSA. Despite these data, to our knowledge, there are no studies that specifically examine the association between the presence of cytokines and surgical complications. The present investigation may be helpful for future studies looking at this relationship.Inflammation has recently been emphasized as a component of the CNS manifestations of OSA as well, including generalized cognitive deficits and post-operative delirium. It is possible that intermittent hypoxia leads to CNS inflammation/activation of microglia (as has been shown in in vitro studies), which, together with blood-brain barrier (BBB) breakdown (recently shown to be involved in OSA), results in elevated circulating peripheral levels of cytokines. Alternatively (or additionally), there could be direct peripheral activation of systemic macrophages as a consequence of sleep deprivation and the cortisol/stress response to this condition. In any event, to date, there are no studies exploring the presence or levels of cytokines in the CSF of patients with OSA. In addition to the release of inflammatory cytokines, activation of microglia causes the release of neuroprotective neurotrophins. Alterations in levels of several neurotrophins have been implicated in multiple CNS diseases. For example, in Parkinson's disease, there is a known elevation in cytokines with reduced circulating levels of CSF neurotrophins (BDNF and NGF) and this balance has been posited to underlie some of the symptoms and progression of the disease. BDNF has recently been shown to protect against the development of Alzheimer's disease and dementia, as well as to increase with caloric restriction and physical activity.

Considering OSA is associated with obesity, it is possible that low BDNF may (at least in part) mediate some of the cognitive deficits seen in OSA. Additionally, low BDNF is associated with postoperative delirium in clinical studies. Currently, the role of neurotrophins in OSA remains underinvestigated. Of all the known neurotrophins, only BDNF has been studied in OSA patients, and the results are conflicting, with some studies suggesting reduced levels of serum BDNF and others showing no differences compared to control patients. This may in part be due to the detection methods employed or small sample sizes, and to date, no one has investigated CSF levels of neurotrophins in this patient population. Here we hypothesize that the detrimental effects of circulating cytokines in OSA may be balanced in some patients by beneficial effects exerted by neurotrophins, and that this differential balance may represent: 1) a tool for identifying which patients are at risk for post-operative complications in future studies, i.e., a useful biomarker for stratifying operative risk; 2) a new understanding of the pathophysiology of OSA; and 3) a role for neuroprotective strategies in the management of OSA.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 50 and 84
* Treated and Untreated OSA Patients: Known OSA, diagnosed by polysomnography
* Treated OSA Patients: Known CPAP prescription, dose used nightly, and compliance status
* Controls: No suspicion for OSA, based on STOP-BANG screening score (<3)
* Any patient presenting for knee replacement surgery with prior consent for spinal or combined spinal-epidural anesthesia

Exclusion Criteria:

* Presence of dementia
* Presence of cognitive disease
* Presence of depression, anxiety, or other mood disorder(s)
* Recent oral steroid therapy (within prior 6 months)
* Requirement of stress-dose steroids pre-operatively
* Autoimmune disease
* Neurologic disease
* Controls: Suspected OSA, either disclosed by patient, or by clinical suspicion based on STOP-BANG questionnaire (score ≥ 3)
* Chronic renal disease
* Chronic liver disease
* Traumatic spinal or spinal-epidural placement (i.e., blood-contaminated CSF)
* Alcohol abuse - defined as being diagnosed with alcohol abuse or consuming more than 2 drinks per night, on average
* Use of NSAIDs within 7 days prior to surgery
* Chronic benzodiazepine use (for more than one month)

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kethy M Jules-Elysee, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Practice guidelines for the perioperative management of patients with obstructive sleep apnea: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Anesthesiology. 2014 Feb;120(2):268-86. doi: 10.1097/ALN.0000000000000053. No abstract available. PMID 24346178
- [Background] Aisen PS. Serum brain-derived neurotrophic factor and the risk for dementia. JAMA. 2014 Apr 23-30;311(16):1684-5. doi: 10.1001/jama.2014.3120. No abstract available. PMID 24756518
- [Background] Baessler A, Nadeem R, Harvey M, Madbouly E, Younus A, Sajid H, Naseem J, Asif A, Bawaadam H. Treatment for sleep apnea by continuous positive airway pressure improves levels of inflammatory markers - a meta-analysis. J Inflamm (Lond). 2013 Mar 22;10:13. doi: 10.1186/1476-9255-10-13. eCollection 2013. PMID 23518041
- [Background] Flink BJ, Rivelli SK, Cox EA, White WD, Falcone G, Vail TP, Young CC, Bolognesi MP, Krystal AD, Trzepacz PT, Moon RE, Kwatra MM. Obstructive sleep apnea and incidence of postoperative delirium after elective knee replacement in the nondemented elderly. Anesthesiology. 2012 Apr;116(4):788-96. doi: 10.1097/ALN.0b013e31824b94fc. PMID 22337162
- [Background] Grandi C, Tomasi CD, Fernandes K, Stertz L, Kapczinski F, Quevedo J, Dal-Pizzol F, Ritter C. Brain-derived neurotrophic factor and neuron-specific enolase, but not S100beta, levels are associated to the occurrence of delirium in intensive care unit patients. J Crit Care. 2011 Apr;26(2):133-7. doi: 10.1016/j.jcrc.2010.10.006. Epub 2010 Nov 23. PMID 21106342
- [Background] Lal C, Strange C, Bachman D. Neurocognitive impairment in obstructive sleep apnea. Chest. 2012 Jun;141(6):1601-1610. doi: 10.1378/chest.11-2214. PMID 22670023
- [Background] Lim DC, Pack AI. Obstructive sleep apnea and cognitive impairment: addressing the blood-brain barrier. Sleep Med Rev. 2014 Feb;18(1):35-48. doi: 10.1016/j.smrv.2012.12.003. Epub 2013 Mar 28. PMID 23541562
- [Background] Nakajima K, Kohsaka S. Microglia: neuroprotective and neurotrophic cells in the central nervous system. Curr Drug Targets Cardiovasc Haematol Disord. 2004 Mar;4(1):65-84. doi: 10.2174/1568006043481284. PMID 15032653
- [Background] Nadeem R, Molnar J, Madbouly EM, Nida M, Aggarwal S, Sajid H, Naseem J, Loomba R. Serum inflammatory markers in obstructive sleep apnea: a meta-analysis. J Clin Sleep Med. 2013 Oct 15;9(10):1003-12. doi: 10.5664/jcsm.3070. PMID 24127144
- [Background] Nagatsu T, Mogi M, Ichinose H, Togari A. Changes in cytokines and neurotrophins in Parkinson's disease. J Neural Transm Suppl. 2000;(60):277-90. doi: 10.1007/978-3-7091-6301-6_19. PMID 11205147
- [Background] Panaree B, Chantana M, Wasana S, Chairat N. Effects of obstructive sleep apnea on serum brain-derived neurotrophic factor protein, cortisol, and lipid levels. Sleep Breath. 2011 Dec;15(4):649-56. doi: 10.1007/s11325-010-0415-7. Epub 2010 Sep 24. PMID 20865453
- [Background] Yang Q, Wang Y, Feng J, Cao J, Chen B. Intermittent hypoxia from obstructive sleep apnea may cause neuronal impairment and dysfunction in central nervous system: the potential roles played by microglia. Neuropsychiatr Dis Treat. 2013;9:1077-86. doi: 10.2147/NDT.S49868. Epub 2013 Aug 5. PMID 23950649
- [Background] Wang WH, He GP, Xiao XP, Gu C, Chen HY. Relationship between brain-derived neurotrophic factor and cognitive function of obstructive sleep apnea/hypopnea syndrome patients. Asian Pac J Trop Med. 2012 Nov;5(11):906-10. doi: 10.1016/S1995-7645(12)60169-2. PMID 23146807

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated OSA (CPAP-compliant): Treated OSA patients will have previously been diagnosed with OSA, and are currently CPAP-compliant. CPAP compliance is defined by daily use of a CPAP machine for at least 4 hours. We will determine if patients are CPAP-compliant by looking at their medical records and pre-operative assessments, as well as directly verifying compliance with the patient.
  Intervention: Lumbar Puncture (Standard-of-Care)
  Lumbar Puncture (Standard-of-Care): All study patients will have previously consented to undergo either spinal or spinal-epidural anesthesia. Patients will undergo their planned spinal or combined spinal-epidural placement in the OR. At the time of confirmation of placement of the spinal needle (positive CSF flow), 5 mL CSF will be collected and stored. CSF will be drawn using a standard 25g or 27g needle commonly used for anesthesia. The volume of CSF removed will be replaced with 4 cc local anesthetic (1.5% mepivacaine for spinal anesthesia).
- Untreated OSA (Non-CPAP-compliant): Patients in the untreated OSA group will have previously been diagnosed with OSA, but for some reason do not use a CPAP machine every night. We will determine if patients are CPAP-compliant by looking at their medical records and pre-operative assessments, as well as directly verifying compliance with the patient.
  Intervention: Lumbar Puncture (Standard-of-Care)
  Lumbar Puncture (Standard-of-Care): All study patients will have previously consented to undergo either spinal or spinal-epidural anesthesia. Patients will undergo their planned spinal or combined spinal-epidural placement in the OR. At the time of confirmation of placement of the spinal needle (positive CSF flow), 5 mL CSF will be collected and stored. CSF will be drawn using a standard 25g or 27g needle commonly used for anesthesia. The volume of CSF removed will be replaced with 4 cc local anesthetic (1.5% mepivacaine for spinal anesthesia).
- Control (No Suspicion of OSA): Patients in the control group will not have previously been diagnosed with OSA, and are currently not at high risk. We will determine overall risk for OSA using the STOP-BANG questionnaire. Patients with a STOP-BANG score <3 are considered to have minimal risk for OSA and will be included in the control group.
  Intervention: Lumbar Puncture (Standard-of-Care)
  Lumbar Puncture (Standard-of-Care): All study patients will have previously consented to undergo either spinal or spinal-epidural anesthesia. Patients will undergo their planned spinal or combined spinal-epidural placement in the OR. At the time of confirmation of placement of the spinal needle (positive CSF flow), 5 mL CSF will be collected and stored. CSF will be drawn using a standard 25g or 27g needle commonly used for anesthesia. The volume of CSF removed will be replaced with 4 cc local anesthetic (1.5% mepivacaine for spinal anesthesia).
Period: Overall Study
Arm/Group | Treated OSA (CPAP-compliant) | Untreated OSA (Non-CPAP-compliant) | Control (No Suspicion of OSA)
Started (1/19/2015) | 16 | 15 | 19
Completed (11/15/16) | 12 | 12 | 13
Not Completed | 4 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treated OSA (CPAP-compliant) | Untreated OSA (Non-CPAP-compliant) | Control (No Suspicion of OSA) | Total
Number analyzed (Participants) | 16 | 15 | 19 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 9 | 5 | 20
  >=65 years | 10 | 6 | 14 | 30
Age, Continuous [Mean (Full Range); unit: years] — Population: Not all participants analyzed fall onto the same range of age
  years | 67.81 [56 to 78] | 63.066 [54 to 72] | 71.68 [51 to 83] | 67.86 [51 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 15 | 29
  Male | 8 | 9 | 4 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 15 | 19 | 50

OUTCOME MEASURES:

1. Primary Outcome: Serum IL-6 (Interleukin 6) Levels
Description: The primary outcome, the levels of cytokine IL-6 in serum of OSA-treated, OSA-untreated and control patients presenting for knee replacement surgery with planned spinal or combined spinal-epidural anesthesia.
Time Frame: Intraoperatively - Pre-Incision
Population: The samples have been collected but the assays have not been performed due to the integrity of the samples.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treated OSA (CPAP-compliant) | Untreated OSA (Non-CPAP-compliant) | Control (No Suspicion of OSA)
Number analyzed (Participants) | 12 | 12 | 13
pg/mL | NA (NA) — The samples have been collected but the assays have not been performed due to the integrity of the samples. | NA (NA) — The samples have been collected but the assays have not been performed due to the integrity of the samples. | NA (NA) — The samples have been collected but the assays have not been performed due to the integrity of the samples.

2. Secondary Outcome: Serum and CSF (Cerebrospinal Fluid) Levels of the Cytokines TNF-alpha (Tumor Necrosis Factor) , IL-6, IL-8, IL-10 (Interleukin)
Description: Biological samples were collected, but not analyzed for the presence and levels of particular cytokines (TNF-alpha, IL-6, IL-8, IL-10) and neurotrophins (BDNF(brain-derived neurotrophic factor), β-NGF (nerve growth factor)) due to the integrity of the samples.
Time Frame: Intraoperatively - Pre-Incision
Reporting Status: Not Posted

3. Secondary Outcome: Serum and CSF Levels of the Neurotrophins BDNF, IFN-gamma (Interferon Gamma)
Description: CSF (cerebrospinal fluid) was planned to be screened for the differential expression of proteins.The samples have been collected, but the assays have not been performed due to the integrity of the samples.
Time Frame: Intraoperatively - Pre-Incision
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants With Respiratory, Cardiac, and/or CNS (Central Nervous System) Complications
Description: We will look at the incidence of respiratory complications (hypoxia; need for respiratory intervention), cardiac complications (MI/ACS or arrhythmias) and CNS (central nervous system) complications (delirium, TIA or CVA). Parameters will be scored for presence or absence over the entire length of stay.
Time Frame: Throughout hospital stay, or an average of 1 week.
Measure: Number; unit: participants
Arm/Group | Treated OSA (CPAP-compliant) | Untreated OSA (Non-CPAP-compliant) | Control (No Suspicion of OSA)
Number analyzed (Participants) | 12 | 12 | 13
participants
  Need for nasal airway | 2 | 5 | 0
  Need for oral airway/airway adjunct | 4 | 4 | 0
  Need for continuous chin lifts | 7 | 8 | 0
  Need for intubation | 0 | 1 | 0
  Need for mechanical ventilation | 2 | 0 | 0

5. Secondary Outcome: Incidence of Intraoperative Obstructive Respiratory Events
Description: Incidences of intraoperative obstructive respiratory events will be collected perioperatively in the operating room by the anesthesiologist
Time Frame: Throughout hospital stay, or an average of 1 week.
Measure: Number; unit: participants
Arm/Group | Treated OSA (CPAP-compliant) | Untreated OSA (Non-CPAP-compliant) | Control (No Suspicion of OSA)
Number analyzed (Participants) | 12 | 12 | 13
participants
  Apneic events | 8 | 9 | 0
  Hypoapnea | 2 | 1 | 2

6. Secondary Outcome: Levels of Blood Oxygen Saturation
Description: Levels of blood oxygen saturation will be measured via arterial blood gas levels. These will be drawn as standard-of-care.
Time Frame: Throughout stay in the recovery unit, or an average of 1-2 days.
Reporting Status: Not Posted

7. Secondary Outcome: Length of Stay in the Recovery Unit
Description: Levels of blood oxygen saturation throughout the length of stay in the recovery unit will be measured via arterial blood gas levels, found in the patient's electronic medical record
Time Frame: Throughout stay in the recovery unit, or an average of 1-2 days.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Treated OSA (CPAP-compliant) | Untreated OSA (Non-CPAP-compliant) | Control (No Suspicion of OSA)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes